CLINICAL TRIAL: NCT00645021
Title: A Phase 1, Open-Label, Parallel Group, Multiple-Dose Study To Evaluate The Pharmacokinetics, Safety And Toleration Of CP-945,598 Administered To Subjects With Impaired And Normal Hepatic Function
Brief Title: Study Examining The Effect Of Hepatic Impairment On Safety, Toleration And How The Body Processes An Experimental Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5351029
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2008-11

CONDITIONS: Obesity; Hepatic Insufficiency
MeSH Terms: conditions — Obesity; Hepatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild hepatic function (Experimental)
  Interventions: Drug: CP-945,598
- Moderate hepatic function (Experimental)
  Interventions: Drug: CP-945,598
- Normal hepatic function (Experimental)
  Interventions: Drug: CP-945,598

INTERVENTIONS:
Drug: CP-945,598 — Administration of CP-945,598 in subjects with mild hepatic function
  Arms: Mild hepatic function
Drug: CP-945,598 — Administration of CP-945,598 in subjects with moderate hepatic function
  Arms: Moderate hepatic function
Drug: CP-945,598 — Administration of CP-945,598 in subjects with normal hepatic function
  Arms: Normal hepatic function

SUMMARY:
CP-945,598 is eliminated following extensive metabolism. Decrease hepatic function can affect its elimination from the body via metabolism. This study will therefore compare the pharmacokinetics (time course of drug concentrations in the body), safety, and tolerability of CP-945,598 in patients with mild and moderate hepatic impairment and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy:Matched for age (± 5 years), weight (± 10 kg), and gender (±2 subjects per gender)
* Subjects with hepatic disease: 1. mild impairment (child-pugh score 5-6), moderate (child-pugh score 7-9). 2. stable hepatic disease: no changes in the last 30 days. 3. stable dose of medication and/or treatment.

Exclusion Criteria:

* All subjects: Non-prescribed use of drugs of abuse/recreational drugs; recent treatment with experimental drugs or herbal experiments; ECG and blood pressure falling outside of protocol-specified limits; history of regular tobacco use exceeding protocol-specified limits
* Normal subjects: medically important health conditions; recent use of prescription or non-prescription medications; history of regular alcohol use exceeding protocol-specified limits
* Subjects with hepatic disease: child-puge score greater than 9; hepatic carcinoma and hepatorenal syndrome;Undergone porta-caval shunt surgery; History of GI hemorrhage due to esophageal varices or peptic ulcers less than 1 month prior to study entry; significant hepatic encephalopathy; severe ascites and/or pleural effusion; Positive blood alcohol test/alcohol breathalyzer at screening or on Day 0.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Measurement of drug and metabolite concentrations in serum collected at various times over 24 hour dosing interval on Days 1 and 14, before daily dose on days 5-7, 13, following stopping of drug treatment on days 15-18, 21, 28, and 35 | 14 days

SECONDARY OUTCOMES:
Safety laboratory tests (chemistry, hematology, urinalysis) on days 0, 7, 15, 35 | 14 days
Adverse event monitoring throughout duration of the study | 14 days
Vital signs (blood pressure, heart rate and respiratory rate) on days 1, 7, and 14 | 14 days
ECGs on Days 1, 7, and 14 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5351029&StudyName=Study%20Examining%20The%20Effect%20Of%20Hepatic%20Impairment%20On%20Safety%2C%20Toleration%20And%20How%20The%20Body%20Processes%20An%20Experimental%20Drug